CLINICAL TRIAL: NCT06882330
Title: Neural Mechanisms of Dialectical Behavioral Therapy in Patients with Borderline Personality Disorder
Acronym: NeuroDBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masarykova Univerzita (Other)
Collaborators: Brno University Hospital (Other); Masaryk University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU20-04-00410
Record Dates: First submitted 2025-02-28; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Borderline Personality Disorder
Keywords: Dialectical behavior therapy; Borderline personality disorder; Therapy effectiveness
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- BPD-DBT group - patients undergoing DBT program. (Experimental): Patients with BPD undergoing Dialectical behavioral therapy (DBT) program with all the standard DBT modules (individual therapy 1 hour per week, skill groups 1.5 hours twice per week, phone coaching as needed, and consultation team 1.5 hours per week). The program lasts a total of 24 weeks in total including two 12-week runs of skills training. Four individual pretreatment sessions precede the program before the start of the main program part.
  Interventions: Behavioral: Dialectical behavior therapy
- BPD-C group - patients undergoing treatment as usual (TAU) (No Intervention): Patients with BPD who are on the waiting list and who receive treatment as usual (typically standard individual psychotherapy not specifically focused on BPD treatment and/or psychiatric treatment).
- HC group: healthy controls (No Intervention): Healthy controls matched to the BPD-DBT group for age and education. Participants without mental health problems and/or a history of self-harm or suicidal behavior. This group receives no psychotherapy or psychiatric treatment.

INTERVENTIONS:
Behavioral: Dialectical behavior therapy — A complex psychotherapy program for patients with borderline personality disorder.
  Arms: BPD-DBT group - patients undergoing DBT program.

SUMMARY:
This research examines the behavioral and neural mechanisms of dialectical behavior therapy (DBT) effect in patients with borderline personality disorder (BPD).

DETAILED DESCRIPTION:
This project aims to evaluate the behavioral and neural mechanisms of dialectical behavior therapy (DBT) effect in patients with borderline personality disorder (BPD). The project includes three subject groups: patients with BPD undergoing the DBT program (BPD-DBT), control patients with BPD on the waiting list for the program (BPD-control), and healthy controls (HC). Patients in the BPD-DBT group undergo a 24-week DBT program in an outpatient setting. All participants undergo a test battery comprising of self-report measures, clinical evaluation and fMRI and EEG measurement in the week before the DBT program beginning (T1), after 24 weeks (follow-up, T3), and at 24 weeks after T3 (follow-up, T4). The BPD-DBT group undergoes another assessment at T2 (after 12 weeks) to monitor selected symptoms during the DBT program by a short set of questionnaires.

ELIGIBILITY:
BPD-DBT group:

Inclusion Criteria:

* diagnosis of borderline personality disorder according to Diagnostic and Statistical Manual 5th Edition (DSM-5) criteria (rated by Structured Clinical Interview for DSM-5 for Personality Disorders, BPD section)
* minimum age 16, informed consent of the patient
* informed consent of patient's legal representative in case of patients under age 18
* more than one self-injury incident and/or suicidal attempt in the past six months

Exclusion Criteria:

* neurological disorder
* comorbid affective disorder or schizophrenia-related disorder
* intelligence quotient<70
* contraindications for MRI measurement
* pregnancy
* body mass index under 15

BPD-C group:

Inclusion Criteria:

* diagnosis of borderline personality disorder according to Diagnostic and Statistical Manual 5th Edition (DSM-5) criteria (rated by Structured Clinical Interview for DSM-5 for Personality Disorders, BPD section)
* minimum age 16, informed consent of the patient
* informed consent of patient's legal representative in case of patients under age 18
* more than one self-injury incident and/or suicidal attempt in the past six months

Exclusion Criteria:

* completing a DBT program or attending DBT-based therapy
* neurological disorder
* comorbid affective disorder or schizophrenia-related disorder
* intelligence quotient<70
* contraindications for MRI measurement
* pregnancy
* body mass index under 15

HC group:

Inclusion criteria:

* minimum age 16, informed consent of the patient
* informed consent of patient's legal representative in case of patients under age 18

Exclusion criteria:

* mental health problems
* history of self-injury or/and suicidal attempt
* neurological disorder
* intelligence quotient<70
* contraindications for MRI measurement
* pregnancy
* body mass index under 15

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Decrease of borderline symptoms | From baseline (T1), a second assessment takes place after 12 weeks (T2), the third assessment takes place 12 weeks after T2 (T3), and the fourth assessment takes place 24 weeks after T3 (T4).
  significant decrease of symptoms measured by Borderline Symptoms List-23
Decrease of self-injury incidents and suicidal attempts | From baseline (T1), the third assessment takes place 24 weeks after T1 (T3), and the fourth assessment takes place 24 weeks after T3 (T4). The second assessment (T2) is not included in this outcome measure.
  significant decrease of self-injury incidents and suicidal attempts assessed by semi-structured interview Lifetime - Suicide Attempt Self-Injury Count

SECONDARY OUTCOMES:
Decrease in the number of days spent in the hospital | From baseline (T1), the third assessment takes place 24 weeks after T1 (T3), and the fourth assessment takes place 24 weeks after T3 (T4). The second assessment (T2) is not included in this outcome measure.
  significant decrease of days spent in the hospital assessed by semi-structured interview -Treatment History Interview
Ecological momentary assessment of emotional variability | From baseline (T1), the third assessment takes place 24 weeks after T1 (T3), and the fourth assessment takes place 24 weeks after T3 (T4). The second assessment (T2) is not included in this outcome measure.
  EMA assesses respondents' emotions in their natural environment. They complete short questionnaires every hour from 9 AM to 9 PM for two days. First, they rate their ability to identify their current emotion (0-100). Then, they choose an emotion or select "An emotion I cannot name" / "No emotion." Next, they rate its intensity (0-100). Finally, they rate their control over the emotion and how overwhelming it feels (both 0-100).
Increase in reasons for living | From baseline (T1), a second assessment takes place after 12 weeks (T2), the third assessment takes place 12 weeks after T2 (T3), and the fourth assessment takes place 24 weeks after T3 (T4).
  significant increase in reasons for living measured by Brief Reasons for Living Inventory 10
Decrease of impulsivity | From baseline (T1), a second assessment takes place after 12 weeks (T2), the third assessment takes place 12 weeks after T2 (T3), and the fourth assessment takes place 24 weeks after T3 (T4).
  significant decrease of impulsivity measured by UPPS-P questionnaire
Increase of mindfulness | From baseline (T1), a second assessment takes place after 12 weeks (T2), the third assessment takes place 12 weeks after T2 (T3), and the fourth assessment takes place 24 weeks after T3 (T4).
  sifnigicant increase of mindfulness measured by Five Facet Mindfulness Questionnaire
Decrease of rejection sensitivity | From baseline (T1), a second assessment takes place after 12 weeks (T2), the third assessment takes place 12 weeks after T2 (T3), and the fourth assessment takes place 24 weeks after T3 (T4).
  significant decrease of rejection sensitivity measured by Rejection Sensitivity RS-Adult questionnaire
Decrease of dissociation symptoms | From baseline (T1), a second assessment takes place after 12 weeks (T2), the third assessment takes place 12 weeks after T2 (T3), and the fourth assessment takes place 24 weeks after T3 (T4).
  significant decrease of dissociation symptoms measured by Multiscale Dissociation Inventory
Decrease of anxiety | From baseline (T1), a second assessment takes place after 12 weeks (T2), the third assessment takes place 12 weeks after T2 (T3), and the fourth assessment takes place 24 weeks after T3 (T4).
  significant decrease of anxiety symptoms measured by Beck Anxiety Inventory
Decrease of depression ranking | From baseline (T1), a second assessment takes place after 12 weeks (T2), the third assessment takes place 12 weeks after T2 (T3), and the fourth assessment takes place 24 weeks after T3 (T4).
  significant decrease of depression symptoms measured by Beck Depression Inventory II, and MADRS clinical rating
Increase of emotion regulation | From baseline (T1), a second assessment takes place after 12 weeks (T2), the third assessment takes place 12 weeks after T2 (T3), and the fourth assessment takes place 24 weeks after T3 (T4).
  significant increase of emotion regulation measured by Difficulties in emotion regulation scale, and ecological momentary assessment
Changes in fMRI neural activity during "Faces task" | From baseline (T1), the third assessment takes place 24 weeks after T1 (T3), and the fourth assessment takes place 24 weeks after T3 (T4). The second assessment (T2) is not included in this outcome measure.
  Significant changes in fMRI neural activity during the "Faces task". During the task, participants view images of faces expressing negative emotions or scrambled versions of the same images as a neutral control. The task is presented in pseudorandomized blocks, with each face displayed for a fixed duration. To maintain attention, participants respond based on the basis of face gender or frame color.
Changes in fMRI neural activity during fMRI neurofeedback | From baseline (T1), the third assessment takes place 24 weeks after T1 (T3), and the fourth assessment takes place 24 weeks after T3 (T4). The second assessment (T2) is not included in this outcome measure.
  fMRI neurofeedback is used to measure changes in fMRI neural activity. During fMRI neurofeedback, patients try to regulate their emotions according to the direction of the arrows (up or down). They receive feedback on how well they are regulating their emotions through a colour scale.
Changes in fMRI neural activity during Cyberball task | From baseline (T1), the third assessment takes place 24 weeks after T1 (T3), and the fourth assessment takes place 24 weeks after T3 (T4). The second assessment (T2) is not included in this outcome measure.
  The Cyberball task is used to measure changes in fMRI neural activity. Participants play a virtual ball-tossing game, believing they are interacting with two other players, though the game is pre-programmed. They control a hand on the screen to pass the ball, while the co-players are represented by animated figures with names and photographs to enhance ecological validity. There are three conditions: inclusion, exclusion, and overinclusion.
Changes in frontal asymmetry during social exclusion measured by EEG | From baseline (T1), the third assessment takes place 24 weeks after T1 (T3), and the fourth assessment takes place 24 weeks after T3 (T4). The second assessment (T2) is not included in this outcome measure.
  EEG is used to assess changes in frontal asymmetry during Cyberball task in fMRI. Frontal asymmetry: EEG alpha power localized in frontal scalp electrodes and differences between left and right hemisphere.
Changes in ECG during fMRI | From baseline (T1), the third assessment takes place 24 weeks after T1 (T3), and the fourth assessment takes place 24 weeks after T3 (T4). The second assessment (T2) is not included in this outcome measure.
  The Brain Products EEG/ExG system is used to assess heart rate variability. Heart rate variability: Mean R-R interval and standard deviation of R-R intervals evaluated in whole fMRI measurement in standard heart beats removing abnormal beats. R peaks detection performed in one channel recording localized on the chest.
Changes in skin conductance during fMRI | From baseline (T1), the third assessment takes place 24 weeks after T1 (T3), and the fourth assessment takes place 24 weeks after T3 (T4). The second assessment (T2) is not included in this outcome measure.
  The Brain Products EEG/ExG system is used to assess changes in skin conductance and monitor the participant's emotional state during the experimental measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Theiner, Ph.D., Principal Investigator — University Hospital Brno
Locations (1):
- University Hospital Brno and Faculty of Medicine, Masaryk University, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
All IPD in anonymized form will be shared upon reasonable request after approval of principal investigator.
Time Frame: One year after publication of the results.
Access Criteria: Access requests can be submitted by email to Central contact person: Pavla Horká Linhartová.